CLINICAL TRIAL: NCT06521957
Title: The Effectiveness of Cognitive Behavioral Therapy in Improving Psycho-Neuro-Endocrine Factors in Women Following In Vitro Fertilization Program
Brief Title: Effectiveness of CBT in Improving Psycho-Neuro-Endocrine Factors in Women Following In Vitro Fertilization Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Principal Investigator, Feranindhya Agiananda, Staff of Psychiatry Department, Head of Consultation-Liaison Psychiatry Division, Fakultas Kedokteran Universitas Indonesia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ND308/UN2.F1/ETIK/PPM0002/2023
Record Dates: First submitted 2024-07-17; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Cognitive Behavioral Therapy; Hormone Disturbance; In Vitro Fertilization
Keywords: Cognitive Behavioral Therapy; Psycho-Neuro-Endocrine; In Vitro Fertilization
MeSH Terms: conditions — Endocrine System Diseases | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy (Experimental): Structured, short-term psychological treatment in the field of cognition that aims to shape adaptive thoughts and behavior.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Treatment As Usual (No Intervention): Administration of information and education regarding in vitro fertilization according to each patient's needs and current stage of treatment.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Cognitive Behavioral Therapy
  Arms: Cognitive Behavioral Therapy

SUMMARY:
The goal of this clinical trial is to learn if Cognitive Behavioral Therapy (CBT) can improve psychological, neurological, and hormonal aspects in women undergoing In Vitro Fertilization (IVF). The main questions it aims to answer are:

* Is CBT effective in improving psychological aspects (anxiety, depression, and coping mechanism) in women undergoing IVF?
* Is CBT effective in improving neuroendocrine aspects (cortisol levels, neuroepinephrine levels, free trioodothyronine levels) in women underoing IVF?

Researchers will compare CBT to no intervention to see if CBT is effective in improving psychoneuroendocrine aspects.

DETAILED DESCRIPTION:
Participants will

* attend 8 appointments once a week, during which they will be given CBT or no intervention
* have their anxiety score, depression score, and dominant coping mechanism assessed before the first appointment and during appointment 3, 6, and 8
* have their cortisol levels, norepinephrine levels, and free triiodothyronine levels assessed before the first appointment and during appointment 3, 6, and 8

ELIGIBILITY:
Inclusion Criteria:

* Women with primary infertility
* Aged 25-42 at the start of the study
* Willing to participate in the study and willing to sign informed consent form
* Minimum education of high school, able to read, write and understand Bahasa Indonesia

Exclusion Criteria:

* Having one or multiple psychotic disorder(s)

Ages: 25 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in anxiety score | Baseline (1 month before IVF program begins/1 week before pre-IVF counselling begins), interim assessments (at the start of IVF program, at 3 weeks of IVF program, and at 5 weeks of IVF program).
  Hamilton Anxiety Rating Scale (HAM-A), Indonesian version, with minimum score of 0 and maximum score of 56. A score of 0-7 indicates no or minimum anxiety; a score of 8-14 indicates mild anxiety; a score of 15-23 indicates moderate anxiety; and a score of 24 and more indicates severe anxiety. Lower score indicates a better outcome.
Improvement in depression score | Baseline (1 month before IVF program begins/1 week before pre-IVF counselling begins), interim assessments (at the start of IVF program, at 3 weeks of IVF program, and at 5 weeks of IVF program).
  Hamilton Depression Rating Scale (HAM-D), Indonesian version, with minimum score of 0 and maximum score of 52. A score of 0-7 indicates no or minimum depression; a score of 8-16 indicates mild depression; a score of 17-23 indicates moderate depression; and a score of 24 and more indicates severe depression. Lower score indicates a better outcome.
Improvement in coping mechanism | Baseline (1 month before IVF program begins/1 week before pre-IVF counselling begins), interim assessments (at the start of IVF program, at 3 weeks of IVF program, and at 5 weeks of IVF program).
  Coping Orientation to the Problem Experienced (COPE), Indonesian version, divided into 2 scales: adaptive coping (active, acceptance, religious) and maladaptive coping (emotion-focused, avoidance), comprising of 61 questions in total. Shift from dominantly maladaptive coping to adaptive coping indicates a better outcome.
Improvement in cortisol levels | Baseline (1 month before IVF program begins/1 week before pre-IVF counselling begins), interim assessments (at the start of IVF program, at 3 weeks of IVF program, and at 5 weeks of IVF program).
  Blood samples are taken from the participants, of which Hormonal Assay test is then performed. 10-20 µg/dl indicates normal range, and lower levels indicate a better outcome.
Improvement in norepinephrine levels | Baseline (1 month before IVF program begins/1 week before pre-IVF counselling begins), interim assessments (at the start of IVF program, at 3 weeks of IVF program, and at 5 weeks of IVF program).
  Blood samples are taken from the participants, of which Hormonal Assay test is then performed. 70-750 pg/dl indicates normal range, and lower levels indicate a better outcome.
Improvement in free triiodothyronine levels | Baseline (1 month before IVF program begins/1 week before pre-IVF counselling begins), interim assessments (at the start of IVF program, at 3 weeks of IVF program, and at 5 weeks of IVF program).
  Blood samples are taken from the participants, of which Hormonal Assay test is then performed. 2.6 - 4.8 pg/ml indicates normal range.

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Toufexis D, Rivarola MA, Lara H, Viau V. Stress and the reproductive axis. J Neuroendocrinol. 2014 Sep;26(9):573-86. doi: 10.1111/jne.12179. PMID 25040027
- [Background] An Y, Sun Z, Li L, Zhang Y, Ji H. Relationship between psychological stress and reproductive outcome in women undergoing in vitro fertilization treatment: psychological and neurohormonal assessment. J Assist Reprod Genet. 2013 Jan;30(1):35-41. doi: 10.1007/s10815-012-9904-x. Epub 2012 Dec 5. PMID 23212833
- [Result] Schliep KC, Mumford SL, Vladutiu CJ, Ahrens KA, Perkins NJ, Sjaarda LA, Kissell KA, Prasad A, Wactawski-Wende J, Schisterman EF. Perceived stress, reproductive hormones, and ovulatory function: a prospective cohort study. Epidemiology. 2015 Mar;26(2):177-84. doi: 10.1097/EDE.0000000000000238. PMID 25643098